CLINICAL TRIAL: NCT03694262
Title: An Open Label, Non-Randomized Multisite Phase II Trial Combining Bevacizumab, Atezolizumab and Rucaparib for the Treatment of Previously Treated Recurrent and Progressive Endometrial Carcinoma
Brief Title: The EndoBARR Trial (Endometrial Bevacizumab, Atezolizumab, Rucaparib)
Acronym: EndoBARR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Genentech, Inc. (Industry); Clovis Oncology, Inc. (Industry)
Responsible Party: Principal Investigator, William Bradley, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EndoBARR
Record Dates: First submitted 2018-09-26; First posted 2018-10-03 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Endometrial Cancer; Uterine Carcinosarcoma
Keywords: recurrent endometrial cancer; Bevacizumab; Atezolizumab; Rucaparib
MeSH Terms: conditions — Endometrial Neoplasms | interventions — rucaparib; Bevacizumab; atezolizumab

STUDY DESIGN:
Intervention Model Description: Cycle length = 21 days Atezolizumab 1,200mg IV on day 1 Bevacizumab 15mg/kg IV on day 1 Rucaparib 600mg orally twice daily by continuous dosing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Cycle length = 21 days Atezolizumab 1,200mg IV on day 1 Bevacizumab 15mg/kg IV on day 1 Rucaparib 600mg orally twice daily by continuous dosing
  Interventions: Drug: Rucaparib; Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Rucaparib — Rucaparib 600mg orally twice daily by continuous dosing
  Other Names: Rubraca
Drug: Bevacizumab — 15mg/kg IV on day 1 of every cycle
  Other Names: Avastin
Drug: Atezolizumab — 1,200mg IV on day 1 of every cycle
  Other Names: Tecentriq

SUMMARY:
To demonstrate the efficacy and safety of the combination of rucaparib, bevacizumab and atezolizumab in recurrent, progressive endometrial carcinoma.

DETAILED DESCRIPTION:
The combination of the three proposed agents offers the opportunity to explore synergistic relationships between antiangiogenic and immunotherapy and antiangiogenic and PARPi. Increasing genetic instability by PARPi and double-strand breaks may lead to a proinflammatory state that would enhance the activity of immunotherapy, leading to synergistic response in a category of solid tumors that lack active therapy. It is expected that increased double-strand breaks may lead to increased expression of immunogenic antigens, increasing the effect of anti-PD-L1 therapy. Phase I data combining the PD-L1 inhibitor durvalamab with either olaparib or cediranib showed good tolerability and evidence of response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have recurrent or persistent/progressive endometrial carcinoma, which is refractory to curative therapy or established treatments. Histologic confirmation of the original primary tumor is required. Stained slides of either the primary or recurrent tumor are required. If primary FFPE samples are not available, a biopsy demonstrating recurrent disease must be obtained. Pathologic Slides/Blocks will be reviewed at the primary site for confirmation.
2. Patients with the following histologic epithelial cell types are eligible: Endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, transitional cell carcinoma and uterine carcinosarcoma (MMT).
3. Patients must have had one prior chemotherapeutic regimen for management of endometrial carcinoma. Chemotherapy administered in conjunction with primary radiation as a radio-sensitizer WILL be counted as a chemotherapy regimen. Patients may have had, but are not required to have received, a second chemotherapeutic regimen for recurrent disease.
4. All patients must have measurable disease, as defined by RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each target lesion must be ≥ 10 mm when measured by

   CT or MRI. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI.
5. Patients may be enrolled if they do not have a target lesion (>= 10 mm lesion or >=15 mm lymph node), if they have measurable disease. This is defined by RECIST 1.1 as a suspicious lesion <10mm or a lymph node >=10mm but <15mm.
6. Patients must have an EGOG Performance Status of 0, 1.
7. Recovery from effects of recent surgery, radiotherapy, or chemotherapy
8. Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated UTI).
9. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration.
10. Any other prior therapy directed at the malignant tumor, including chemotherapy and immunologic agents, must be discontinued at least three weeks prior to first cycle of treatment.
11. Any prior radiation therapy must be completed at least four weeks prior to first cycle of treatment.
12. Prior hormonal therapy is allowed. There is no limit on the number of prior hormonal therapies allowed. Hormonal therapy will not be counted as a line of therapy for purposes of this trial.
13. Patients must have a urine protein of 2+ on dipstick. If dipstick is >2+, 24-hour urine protein must be obtained and should be < 1g for patient to be eligible.
14. Patients must have signed an approved informed consent and authorization permitting release of personal health information for study purposes.
15. Patients must meet pre-entry requirements, as specified in section 5.
16. Patients of childbearing potential must agree to use an accepted and effective nonhormonal method of contraception i.e., double-barrier method (e.g., condom plus diaphragm) from the time of signing the informed consent through six months after last dose of study drug.
17. Patients 18 years of age or greater.
18. Be willing to provide tissue from the primary surgical resection (paraffin block).
19. Must have laboratory values in the below ranges:

System Laboratory Value Endocrine Thyroid function testing (TSH) 0.350 - 5.500 ulU/mL (Or within institutional labarotory range).

Free T4/Total T3 If TSH is outside of laboratory range and subject is clinically euthyroid, enrollment may occur if Free T4/Total T3 are in normal range by local lab values Hematological

System Laboratory Value Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Renal Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR

≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR

≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.

4.2 Exclusion Criteria

1. Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of the other malignancy being present within the last two years. Patients with Ductal Carcinoma in situ (DCIS) of the breast in the prior two years may be enrolled on study if the treatment required no chemotherapy or radiation. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
2. Patients must not have had exposure to Bevacizumab, PARPi, or immunotherapy. Patients may have had exposure to anti-angiogentic therapy provided it was not Bevacizumab.
3. Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer within the last three years are excluded. Prior radiation for localized cancer of the breast, head and neck or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
4. Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of endometrial cancer within the last three years are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than two years prior to registration, and that the patient remains free of recurrent or metastatic disease.
5. Inability to tolerate an oral medication or keep pills down.
6. Patients who are pregnant or nursing.
7. Patients with a complete bowel obstruction; recent (within six months) history of fistula, intraabdominal abscess or bowel perforation; subjects requiring total parenteral nutrition or parenteral hydration.
8. Has a current diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within seven days prior to the first dose of trial treatment.
9. Patients with history or evidence upon physical examination of CNS disease, including brain tumor, seizures not controlled with standard medical therapy or any brain metastases.
10. Patients with clinically significant cardiovascular disease. This includes:

    * Myocardial infarction or unstable angina within 12 months of the first date of study treatment.
    * New York Heart Association (NYHA) Class II or greater congestive heart failure (Appendix I).
    * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation) or cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication).
    * Grade 2 or greater peripheral vascular disease.
    * Cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of study treatment.
    * History of arterial ischemia or thrombus.
11. Patients with uncontrolled hypertension defined as systolic > 150 mm Hg or diastolic > 90 mm Hg. The use of antihypertensive medications to control hypertension is permitted.
12. Patients who have undergone major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of study treatment or who have a major surgical procedure anticipated during the course of the study. Laparoscopic biopsy is acceptable and will not require a delay in study treatment.
13. Patients with serious nonhealing wound, ulcer (including gastrointestinal) or bone fracture.
14. Patients with any condition, which in the investigator's opinion, makes the patient unsuitable for study participation.
15. Patients not available for follow-up assessments.
16. Patients with known sensitivity to any of the products to be administered during dosing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2026-01-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William Bradley, MD, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - Mount Sinai, New York, New York
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Froedtert Lutheran Memorial Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aghajanian, C., Filiaci, V.L., Dizon, D.S., Carlson, J., Powell, M.A., Secord, A.A., Tewari, K.S., Bender, D., O'Malley, D.M., Stuckey, A., et al. (2015). A randomized phase II study of paclitaxel/carboplatin/bevacizumab, paclitaxel/carboplatin/temsirolimus and ixabepilone/carboplatin/bevacizumab as initial therapy for measurable stage III or IVA, stage IVB or recurrent endometrial cancer, GOG-86P. Journal of Clinical Oncology 33, 5500-5500.
- [Result] Aghajanian C, Sill MW, Darcy KM, Greer B, McMeekin DS, Rose PG, Rotmensch J, Barnes MN, Hanjani P, Leslie KK. Phase II trial of bevacizumab in recurrent or persistent endometrial cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2011 Jun 1;29(16):2259-65. doi: 10.1200/JCO.2010.32.6397. Epub 2011 May 2. PMID 21537039
- [Result] Arielle Lutterman Heeke, T.B., Filipa Lynce, Michael J. Pishvaian, Claudine Isaacs (2017). Prevalence of homologous recombination deficiency among all tumor types. Journal of Clinical Oncology 35.
- [Result] Bhattacharya S, Fyfe G, Gray RJ, Sargent DJ. Role of sensitivity analyses in assessing progression-free survival in late-stage oncology trials. J Clin Oncol. 2009 Dec 10;27(35):5958-64. doi: 10.1200/JCO.2009.22.4329. Epub 2009 Oct 13. PMID 19826121
- [Result] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Result] Carlson MJ, Thiel KW, Leslie KK. Past, present, and future of hormonal therapy in recurrent endometrial cancer. Int J Womens Health. 2014 May 2;6:429-35. doi: 10.2147/IJWH.S40942. eCollection 2014. PMID 24833920
- [Result] Castonguay V, Lheureux S, Welch S, Mackay HJ, Hirte H, Fleming G, Morgan R, Wang L, Blattler C, Ivy PS, Oza AM. A phase II trial of sunitinib in women with metastatic or recurrent endometrial carcinoma: a study of the Princess Margaret, Chicago and California Consortia. Gynecol Oncol. 2014 Aug;134(2):274-80. doi: 10.1016/j.ygyno.2014.05.016. Epub 2014 May 29. PMID 24882554
- [Result] Choueiri TK, Mayer EL, Je Y, Rosenberg JE, Nguyen PL, Azzi GR, Bellmunt J, Burstein HJ, Schutz FA. Congestive heart failure risk in patients with breast cancer treated with bevacizumab. J Clin Oncol. 2011 Feb 20;29(6):632-8. doi: 10.1200/JCO.2010.31.9129. Epub 2011 Jan 4. PMID 21205755
- [Result] Coleman RL, Sill MW, Lankes HA, Fader AN, Finkler NJ, Hoffman JS, Rose PG, Sutton GP, Drescher CW, McMeekin DS, Hu W, Deavers M, Godwin AK, Alpaugh RK, Sood AK. A phase II evaluation of aflibercept in the treatment of recurrent or persistent endometrial cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 Dec;127(3):538-43. doi: 10.1016/j.ygyno.2012.08.020. Epub 2012 Aug 23. PMID 22922531
- [Result] Cosgrove CM, Cohn DE, Hampel H, Frankel WL, Jones D, McElroy JP, Suarez AA, Zhao W, Chen W, Salani R, Copeland LJ, O'Malley DM, Fowler JM, Yilmaz A, Chassen AS, Pearlman R, Goodfellow PJ, Backes FJ. Epigenetic silencing of MLH1 in endometrial cancers is associated with larger tumor volume, increased rate of lymph node positivity and reduced recurrence-free survival. Gynecol Oncol. 2017 Sep;146(3):588-595. doi: 10.1016/j.ygyno.2017.07.003. Epub 2017 Jul 11. PMID 28709704
- [Result] Fleming GF. Second-Line Therapy for Endometrial Cancer: The Need for Better Options. J Clin Oncol. 2015 Nov 1;33(31):3535-40. doi: 10.1200/JCO.2015.61.7225. Epub 2015 Jul 20. No abstract available. Erratum In: J Clin Oncol. 2015 Dec 20;33(36):4316. doi: 10.1200/JCO.2015.65.7080. PMID 26195695
- [Result] Fleming GF, Brunetto VL, Cella D, Look KY, Reid GC, Munkarah AR, Kline R, Burger RA, Goodman A, Burks RT. Phase III trial of doxorubicin plus cisplatin with or without paclitaxel plus filgrastim in advanced endometrial carcinoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2004 Jun 1;22(11):2159-66. doi: 10.1200/JCO.2004.07.184. PMID 15169803
- [Result] Gabrilovich DI, Chen HL, Girgis KR, Cunningham HT, Meny GM, Nadaf S, Kavanaugh D, Carbone DP. Production of vascular endothelial growth factor by human tumors inhibits the functional maturation of dendritic cells. Nat Med. 1996 Oct;2(10):1096-103. doi: 10.1038/nm1096-1096. PMID 8837607
- [Result] Goldberg SB, Narayan A, Kole AJ, Decker RH, Teysir J, Carriero NJ, Lee A, Nemati R, Nath SK, Mane SM, Deng Y, Sukumar N, Zelterman D, Boffa DJ, Politi K, Gettinger SN, Wilson LD, Herbst RS, Patel AA. Early Assessment of Lung Cancer Immunotherapy Response via Circulating Tumor DNA. Clin Cancer Res. 2018 Apr 15;24(8):1872-1880. doi: 10.1158/1078-0432.CCR-17-1341. Epub 2018 Jan 12. PMID 29330207
- [Result] Goodfellow PJ, Billingsley CC, Lankes HA, Ali S, Cohn DE, Broaddus RJ, Ramirez N, Pritchard CC, Hampel H, Chassen AS, Simmons LV, Schmidt AP, Gao F, Brinton LA, Backes F, Landrum LM, Geller MA, DiSilvestro PA, Pearl ML, Lele SB, Powell MA, Zaino RJ, Mutch D. Combined Microsatellite Instability, MLH1 Methylation Analysis, and Immunohistochemistry for Lynch Syndrome Screening in Endometrial Cancers From GOG210: An NRG Oncology and Gynecologic Oncology Group Study. J Clin Oncol. 2015 Dec 20;33(36):4301-8. doi: 10.1200/JCO.2015.63.9518. Epub 2015 Nov 9. PMID 26552419
- [Result] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Result] Heinzerling L, Ott PA, Hodi FS, Husain AN, Tajmir-Riahi A, Tawbi H, Pauschinger M, Gajewski TF, Lipson EJ, Luke JJ. Cardiotoxicity associated with CTLA4 and PD1 blocking immunotherapy. J Immunother Cancer. 2016 Aug 16;4:50. doi: 10.1186/s40425-016-0152-y. eCollection 2016. PMID 27532025
- [Result] Herrmann J, Lerman A, Sandhu NP, Villarraga HR, Mulvagh SL, Kohli M. Evaluation and management of patients with heart disease and cancer: cardio-oncology. Mayo Clin Proc. 2014 Sep;89(9):1287-306. doi: 10.1016/j.mayocp.2014.05.013. PMID 25192616
- [Result] Higuchi T, Flies DB, Marjon NA, Mantia-Smaldone G, Ronner L, Gimotty PA, Adams SF. CTLA-4 Blockade Synergizes Therapeutically with PARP Inhibition in BRCA1-Deficient Ovarian Cancer. Cancer Immunol Res. 2015 Nov;3(11):1257-68. doi: 10.1158/2326-6066.CIR-15-0044. Epub 2015 Jul 2. PMID 26138335
- [Result] Jiao S, Xia W, Yamaguchi H, Wei Y, Chen MK, Hsu JM, Hsu JL, Yu WH, Du Y, Lee HH, Li CW, Chou CK, Lim SO, Chang SS, Litton J, Arun B, Hortobagyi GN, Hung MC. PARP Inhibitor Upregulates PD-L1 Expression and Enhances Cancer-Associated Immunosuppression. Clin Cancer Res. 2017 Jul 15;23(14):3711-3720. doi: 10.1158/1078-0432.CCR-16-3215. Epub 2017 Feb 6. PMID 28167507
- [Result] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Result] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Result] Lee JM, Cimino-Mathews A, Peer CJ, Zimmer A, Lipkowitz S, Annunziata CM, Cao L, Harrell MI, Swisher EM, Houston N, Botesteanu DA, Taube JM, Thompson E, Ogurtsova A, Xu H, Nguyen J, Ho TW, Figg WD, Kohn EC. Safety and Clinical Activity of the Programmed Death-Ligand 1 Inhibitor Durvalumab in Combination With Poly (ADP-Ribose) Polymerase Inhibitor Olaparib or Vascular Endothelial Growth Factor Receptor 1-3 Inhibitor Cediranib in Women's Cancers: A Dose-Escalation, Phase I Study. J Clin Oncol. 2017 Jul 1;35(19):2193-2202. doi: 10.1200/JCO.2016.72.1340. Epub 2017 May 4. PMID 28471727
- [Result] Lincoln S, Blessing JA, Lee RB, Rocereto TF. Activity of paclitaxel as second-line chemotherapy in endometrial carcinoma: a Gynecologic Oncology Group study. Gynecol Oncol. 2003 Mar;88(3):277-81. doi: 10.1016/s0090-8258(02)00068-9. PMID 12648575
- [Result] Liu JF, Barry WT, Birrer M, Lee JM, Buckanovich RJ, Fleming GF, Rimel B, Buss MK, Nattam S, Hurteau J, Luo W, Quy P, Whalen C, Obermayer L, Lee H, Winer EP, Kohn EC, Ivy SP, Matulonis UA. Combination cediranib and olaparib versus olaparib alone for women with recurrent platinum-sensitive ovarian cancer: a randomised phase 2 study. Lancet Oncol. 2014 Oct;15(11):1207-14. doi: 10.1016/S1470-2045(14)70391-2. Epub 2014 Sep 10. PMID 25218906
- [Result] Makker V, Green AK, Wenham RM, Mutch D, Davidson B, Miller DS. New therapies for advanced, recurrent, and metastatic endometrial cancers. Gynecol Oncol Res Pract. 2017 Dec 2;4:19. doi: 10.1186/s40661-017-0056-7. eCollection 2017. PMID 29214032
- [Result] Matson V, Fessler J, Bao R, Chongsuwat T, Zha Y, Alegre ML, Luke JJ, Gajewski TF. The commensal microbiome is associated with anti-PD-1 efficacy in metastatic melanoma patients. Science. 2018 Jan 5;359(6371):104-108. doi: 10.1126/science.aao3290. PMID 29302014
- [Result] McMeekin DS, Tritchler DL, Cohn DE, Mutch DG, Lankes HA, Geller MA, Powell MA, Backes FJ, Landrum LM, Zaino R, Broaddus RD, Ramirez N, Gao F, Ali S, Darcy KM, Pearl ML, DiSilvestro PA, Lele SB, Goodfellow PJ. Clinicopathologic Significance of Mismatch Repair Defects in Endometrial Cancer: An NRG Oncology/Gynecologic Oncology Group Study. J Clin Oncol. 2016 Sep 1;34(25):3062-8. doi: 10.1200/JCO.2016.67.8722. Epub 2016 Jun 20. PMID 27325856
- [Result] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Popescu BA, Waggoner AD. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2016 Apr;29(4):277-314. doi: 10.1016/j.echo.2016.01.011. No abstract available. PMID 27037982
- [Result] Ott PA, Bang YJ, Berton-Rigaud D, Elez E, Pishvaian MJ, Rugo HS, Puzanov I, Mehnert JM, Aung KL, Lopez J, Carrigan M, Saraf S, Chen M, Soria JC. Safety and Antitumor Activity of Pembrolizumab in Advanced Programmed Death Ligand 1-Positive Endometrial Cancer: Results From the KEYNOTE-028 Study. J Clin Oncol. 2017 Aug 1;35(22):2535-2541. doi: 10.1200/JCO.2017.72.5952. Epub 2017 May 10. PMID 28489510
- [Result] Ott PA, Hodi FS, Buchbinder EI. Inhibition of Immune Checkpoints and Vascular Endothelial Growth Factor as Combination Therapy for Metastatic Melanoma: An Overview of Rationale, Preclinical Evidence, and Initial Clinical Data. Front Oncol. 2015 Sep 22;5:202. doi: 10.3389/fonc.2015.00202. eCollection 2015. PMID 26442214
- [Result] Powell MA, Sill MW, Goodfellow PJ, Benbrook DM, Lankes HA, Leslie KK, Jeske Y, Mannel RS, Spillman MA, Lee PS, Hoffman JS, McMeekin DS, Pollock PM. A phase II trial of brivanib in recurrent or persistent endometrial cancer: an NRG Oncology/Gynecologic Oncology Group Study. Gynecol Oncol. 2014 Oct;135(1):38-43. doi: 10.1016/j.ygyno.2014.07.083. Epub 2014 Jul 11. PMID 25019571
- [Result] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Result] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Result] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Result] Thavendiranathan P, Poulin F, Lim KD, Plana JC, Woo A, Marwick TH. Use of myocardial strain imaging by echocardiography for the early detection of cardiotoxicity in patients during and after cancer chemotherapy: a systematic review. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt A):2751-68. doi: 10.1016/j.jacc.2014.01.073. Epub 2014 Apr 2. PMID 24703918
- [Result] Totzeck M, Mincu RI, Rassaf T. Cardiovascular Adverse Events in Patients With Cancer Treated With Bevacizumab: A Meta-Analysis of More Than 20 000 Patients. J Am Heart Assoc. 2017 Aug 10;6(8):e006278. doi: 10.1161/JAHA.117.006278. PMID 28862931
- [Result] Varricchi G, Marone G, Mercurio V, Galdiero MR, Bonaduce D, Tocchetti CG. Immune Checkpoint Inhibitors and Cardiac Toxicity: An Emerging Issue. Curr Med Chem. 2018;25(11):1327-1339. doi: 10.2174/0929867324666170407125017. PMID 28403786

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 30
Treated | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.5 [63 to 73.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — United States of America
  Participants
    United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: To estimate the overall response rate (ORR) of patients with progressive/persistent or recurrent endometrial cancer on study-directed therapy, using the combination of rucaparib, bevacizumab and atezolizumab.
Time Frame: 44 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: To Estimate the Overall Response Rate (ORR) of Patients With Progressive/Persistent or Recurrent Endometrial Cancer on Study-directed Therapy, Using the Combination of Rucaparib, Bevacizumab and Atezolizumab.
Description: overall response rate
Time Frame: Through study completion, up to 3 years. Measured in relation to change from baseline imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 30
Participants | 30

3. Secondary Outcome: Progression Free Survival
Description: Progression-Free Survival (PFS) is defined as the duration of time from date of study entry to time of progression or death, whichever occurs first. The outcome is to estimate the progression free survival (PFS) of patients with progressive/persistent or recurrent endometrial cancer when treated with the combination of rucaparib, bevacizumab and atezolizumab.
Time Frame: 48-60 months
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE V5.0
Description: To determine the nature and degree of toxicity of treatment using the CTCAE v5.0 with this combination in this cohort of patients.
Time Frame: 30-36 months
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Description: Survival is defined as the duration of time from date of study entry to time of death or the date of last contact. The outcome is to estimate the overall survival of patients with persistent or recurrent endometrial cancer, when treated with the combination of rucaparib, bevacizumab and atezolizumab.
Time Frame: 48-60 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Microsatellite Instability (MSI) - Both Genetic and Epigenetic
Description: Measurement of tumor MicroSatellite Instablility (MSI) via both qtPCR (quantitative polymerase chain reaction) and IHC (immunohistochemistry).
Time Frame: 48-60 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Homologus Recombination Deficiency Gene Alterations
Description: Tumor samples will assess for the genes that lead to homologus recombination deficiency.
Time Frame: 48-60 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: PD-L1 Expression in the Tumor
Description: Tumor samples (from initial diagnosis) will have PD-L1 assessed by IHC (immunohistochemistry).
Time Frame: 48-60 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Tumor Mutational Burden
Description: This level will be assessed in primary patient specimens using formalin fixed, paraffin-embedded samples.
Time Frame: 48-60 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Loss of Heterozygosity
Description: Tumor sample will be assessed for loss of heterozygosity
Time Frame: 48-60 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Circulating Tumor DNA
Description: Peripheral blood draw will be assessed for circulating tumor DNA
Time Frame: 48-60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3.5 years
Description: Reporting from sites
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 15/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT03694262/Prot_SAP_002.pdf